CLINICAL TRIAL: NCT04944316
Title: Physicians Committee for Responsible Medicine - a Randomized, Controlled Study of the Effect of a Low-fat, Plant-based Diet on Insulin Requirements in Individuals with Type 1 Diabetes
Brief Title: Effect of a Dietary Intervention on Insulin Requirements in Type 1 Diabetes
Acronym: T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00048903
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-fat, vegan diet (Active Comparator): For a 12-week period, participants will be asked to follow a low-fat, vegan diet which consists of whole grains, vegetables, legumes, and fruits, with no restriction on energy intake. Animal products and added oils will be excluded. In choosing grain products and starchy vegetables (e.g., bread, potatoes), participants will be encouraged to select those retaining their natural fiber and having a glycemic index <70, using tables standardized to a value of 100 for glucose.
  Interventions: Behavioral: Dietary intervention
- Portion-controlled diet (Active Comparator): For a 12-week period, participants will be asked to follow a portion-controlled diet that is compliant with American Diabetes Association (ADA) guidelines. This diet will include individualized diet plans that reduce daily energy intake by 500-1,000 kcal for overweight (body mass index > 25 kg/m2) participants and keep carbohydrate intake reasonably stable over time. It will derive 15-20% from protein, <7% saturated fat, 60-70% carbohydrate and monounsaturated fats and ≤200 mg/day of cholesterol/day.
  Interventions: Behavioral: Dietary intervention

INTERVENTIONS:
Behavioral: Dietary intervention — Low-fat, plant-based diet
  Arms: Low-fat, vegan diet
Behavioral: Dietary intervention — Portion-controlled diet (compliant with ADA guidelines)
  Arms: Portion-controlled diet

SUMMARY:
The purpose of this study is to compare the effects of a low-fat, plant-based dietary intervention and a portion-controlled dietary intervention (compliant with current American Diabetes Association (ADA) guidelines) on the management of type 1 diabetes in adults. The primary outcome measure of this study is insulin requirements (measured as the total daily dose (TDD) of insulin or basal and bolus insulin units injected per day). The study duration is 12 weeks.

DETAILED DESCRIPTION:
Type 1 diabetes is a chronic autoimmune disorder characterized by loss of β-cell mass and function in the pancreas, leading to reduced secretion of insulin and hyperglycemia. The management of type 1 diabetes requires the administration of exogeneous insulin. Total daily dose (TDD) of insulin, a measure of the total amount of exogeneous insulin utilized per day, can be affected by multiple factors including insulin resistance, carbohydrate intake, body weight, and body composition. While the pathogenesis of type 1 diabetes and type 2 diabetes differ, a low-fat, plant-based diet has been shown to reduce insulin resistance, reduce body weight, improve body composition, and improve glycemic control in individuals with type 2 diabetes. A low-fat, plant-based diet has also been shown to improve β-cell function in individuals who are overweight. This finding is consistent with other research that shows that therapies that reduce body fat, or modify the distribution of body fat, improve β-cell function and glucose homeostasis. To date, a low-fat, plant-based diet has never been adequately tested in adults with type 1 diabetes. The purpose of this study is to compare the effects of low-fat, plant-based dietary intervention and a portion-controlled dietary intervention (compliant with current American Diabetes Association (ADA) guidelines) on insulin requirements in adults with type 1 diabetes.

Using a parallel group design, participants with type 1 diabetes will be randomly assigned to follow a low-fat, plant-based diet or a portion-controlled diet (compliant with current ADA guidelines) for 12 weeks. The principal dependent measures of this study are TDD of insulin, hemoglobin A1c (HbA1c), interstitial fluid glucose levels, and 24-hour carbohydrate: insulin ratio. Secondary and tertiary dependent measures include inflammatory biomarkers, blood lipids, body weight, diet quality, diet acceptability, and medication use.

The investigators hypothesize that both the low-fat, plant-based dietary intervention and the portion-controlled dietary intervention will elicit changes in insulin requirements, HbA1c, variability in interstitial glucose levels, insulin sensitivity, and body weight in participants with type 1 diabetes. The investigators further hypothesize that the low-fat, plant-based dietary intervention will confer a more substantial effect on changes in insulin requirements, HbA1c, insulin sensitivity, variability in interstitial glucose levels, and body weight in participants with type 1 diabetes.

ELIGIBILITY:
Inclusion criteria:

1. Type 1 diabetes
2. Men and women ≥ 18 years of age
3. Stable insulin regimen for past 3 months

Exclusion criteria:

1. Type 2 or gestational diabetes
2. Body mass index ≥ 40 kg/m2
3. HbA1c ≥ 12.0%
4. Smoking or drug abuse during the past six months
5. Alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
6. Unstable medical or psychiatric illness
7. Already following a low-fat vegan diet
8. Pregnant or breastfeeding, or plans of pregnancy within the study period
9. Lack of English fluency
10. Unable or unwilling to participate in all components of the study
11. Evidence of an eating disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Total Insulin Dose | Change from week 0 to week 12
  A sum of basal and bolus insulin units (U) injected per day. An average from three (3) days (two (2) workdays and one (1) weekend day) will be utilized.
Glycemic Control | Change from week 0 to week 12
  Hemoglobin A1c (HbA1c), an index of glycemic control, will be utilized.
Glycemic Variability | Change from week 0 to week 12
  Glycemic variability will be assessed through use of a continuous glucose monitoring (CGM) system that will measure the concentration of glucose in the interstitial fluid. Participants will be instructed to wear a CGM (Dexcom g6 Platinum CGM System with an enhanced algorithm, software 505, Dexcom, Inc.) and record its readings at preset increments (after an overnight fast, before each meal, 2 hours after each meal, and before going to bed) daily. Participants will be prompted to submit CGM data to investigators on a weekly basis.
24-hour Carbohydrate to Insulin Ratio | Change from week 0 to week 12
  Calculated as the total number of grams (g) of dietary carbohydrate to total units (U) of insulin administered.

SECONDARY OUTCOMES:
Body Weight | Change from week 0 to week 12
  Change in body weight measured on a calibrated scale.
Concentration of Plasma Lipids | Change from week 0 to week 12
  Change in plasma cholesterol & triglycerides.
High-sensitivity C-reactive Protein (hs-CRP) | Change from week 0 to week 12
  Implemented as a biomarker for absolute cardiovascular disease risk prediction.
Tumor necrosis factor - α (TNF-α) | Change from week 0 to week 12
  Implemented to assess levels of systemic inflammation.
Interleukin (IL) - 1 (IL-1) and interleukin-6 (IL-6) | Change from week 0 to week 12
  Implemented to assess levels of systemic inflammation.
Food costs | 12 weeks
  Food costs will be assessed, using the U.S. Department of Agriculture Thrifty Food Plan, 2021, at baseline and 12 weeks.
Insulin costs | 12 weeks
  Insulin costs will be assessed, using the Federal Supply Schedule (FSS) for insulin prices, at baseline and 12 weeks.

OTHER OUTCOMES:
Medication Use | Change from week 0 to week 12
  Participants will be asked to report changes in their medication use.
Diet Quality | Change from week 0 to week 12
  Dietary intake will be assessed using 3-day dietary records. Participants will be instructed to record all dietary intake for 3 consecutive days, including 2 weekdays and 1 weekend day. Records will be analyzed using Nutrition Data System for Research software version 2018, developed by the Nutrition Coordinating Center (NCC), University of Minnesota, Minneapolis, MN, US.
Diet Acceptability | Change from week 0 to week 12
  The Food Acceptability Questionnaire (FAQ), a self-reported measure, will be implemented to assess the subjective responses (palatability; satisfaction; ease of preparation; financial feasibility; and perceived physical benefits) of participants to their baseline diets and the intervention diet. The FAQ has twelve (12) total questions. Eleven (11) of the questions are scored on a Likert scale (1-7) and one (1) unscored question (physical benefits) will prompt the participant to "check all that apply." A higher FAQ score corresponds with a more positive subjective response.

CONTACTS AND LOCATIONS:
Overall Officials: Hana Kahleova, MD, PhD, Principal Investigator — Physicians Committee for Responsible Medicine
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riccardi G, Rivellese AA, Giacco R. Role of glycemic index and glycemic load in the healthy state, in prediabetes, and in diabetes. Am J Clin Nutr. 2008 Jan;87(1):269S-274S. doi: 10.1093/ajcn/87.1.269S. PMID 18175767
- [Background] Anderson JW, Zeigler JA, Deakins DA, Floore TL, Dillon DW, Wood CL, Oeltgen PR, Whitley RJ. Metabolic effects of high-carbohydrate, high-fiber diets for insulin-dependent diabetic individuals. Am J Clin Nutr. 1991 Nov;54(5):936-43. doi: 10.1093/ajcn/54.5.936. PMID 1659172
- [Background] American Diabetes Association. Standards of Medical Care in Diabetes-2018 Abridged for Primary Care Providers. Clin Diabetes. 2018 Jan;36(1):14-37. doi: 10.2337/cd17-0119. No abstract available. PMID 29382975
- [Background] Pastors JG, Franz MJ, Warshaw H, Daly A, Arnold MS. How effective is medical nutrition therapy in diabetes care? J Am Diet Assoc. 2003 Jul;103(7):827-31. doi: 10.1016/s0002-8223(03)00466-8. No abstract available. PMID 12830019
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Mari A, Tura A, Gastaldelli A, Ferrannini E. Assessing insulin secretion by modeling in multiple-meal tests: role of potentiation. Diabetes. 2002 Feb;51 Suppl 1:S221-6. doi: 10.2337/diabetes.51.2007.s221. PMID 11815483
- [Background] Kahleova H, Mari A, Nofrate V, Matoulek M, Kazdova L, Hill M, Pelikanova T. Improvement in beta-cell function after diet-induced weight loss is associated with decrease in pancreatic polypeptide in subjects with type 2 diabetes. J Diabetes Complications. 2012 Sep-Oct;26(5):442-9. doi: 10.1016/j.jdiacomp.2012.05.003. Epub 2012 Jun 4. PMID 22673566
- [Background] American Dietetic Association; Dietitians of Canada. Position of the American Dietetic Association and Dietitians of Canada: Vegetarian diets. J Am Diet Assoc. 2003 Jun;103(6):748-65. doi: 10.1053/jada.2003.50142. PMID 12778049
- [Background] Barnard ND, Akhtar A, Nicholson A. Factors that facilitate compliance to lower fat intake. Arch Fam Med. 1995 Feb;4(2):153-8. doi: 10.1001/archfami.4.2.153. PMID 7842153
- [Background] Becker MH. The health belief model and personal health behavior. Health Educ Monogr. 1974;2:324-508.
- [Background] Barnard N, Scialli AR, Bertron P, Hurlock D, Edmonds K. Acceptability of a Therapeutic Low-Fat, Vegan Diet in Premenopausal Women. J Nutr Educ. 2000;32(6):314-319. doi:10.1016/S0022-3182(00)70590-5
- [Derived] Kahleova H, Maracine C, Znayenko-Miller T, Kuo S, Herman WH, Holubkov R, Barnard ND. Can a vegan diet help people with type 1 diabetes save on insulin? A secondary analysis of a 12-Week randomized clinical trial. BMC Nutr. 2025 Oct 14;11(1):188. doi: 10.1186/s40795-025-01175-2. PMID 41088465
- [Derived] Kahleova H, Himmelfarb J, Znayenko-Miller T, Jayaraman A, Chiavaroli L, Holubkov R, Barnard ND. Vegan diet, processed foods, and type 1 diabetes: A secondary analysis of a randomized clinical trial. Nutr Metab Cardiovasc Dis. 2025 Nov;35(11):104197. doi: 10.1016/j.numecd.2025.104197. Epub 2025 Jun 13. PMID 40651893
- [Derived] Kahleova H, Fischer I, Smith R, Himmelfarb J, Znayenko-Miller T, Holubkov R, Barnard ND. Plant-based dietary index and body weight in people with type 1 diabetes: a secondary analysis of a randomized clinical trial. Front Nutr. 2025 May 22;12:1605769. doi: 10.3389/fnut.2025.1605769. eCollection 2025. PMID 40474900